CLINICAL TRIAL: NCT04905875
Title: Prone Positioning for Invasively Ventilated Patients With COVID-19: an Interactive, Web-based, Multicenter, Observational Registry
Brief Title: Prone Positioning for Invasively Ventilated Patients With COVID-19 Registry
Acronym: PROVENT-C19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Principal Investigator, Silvia De Rosa, Principal Investigator, St. Bortolo Hospital
Other Study IDs: 22/21
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients with COVID-19: n centres that obtained IRB approval for this prospective study, all critically ill adult patients (>18yrs) undergoing PP - that are homogeneous in terms of both clinical and treatment characteristics - will be prospectively observed.
  Interventions: Procedure: Prone Position

INTERVENTIONS:
Procedure: Prone Position — Every center will prescribe PP in accordance with local practice and local levels of expertise. No variation in treatment prescription and/or treatment solutions will derive from participation in this prospective observational study. Nonetheless, every setting parameter will be recorded in the web-based registry and analyzed a-posteriori to reveal a potential correlation with the patient outcomes.

SUMMARY:
SARS-CoV-2 infection is characterized mainly by moderate/severe pneumonia associated with progressive endothelial damage and coagulopathy. Acute respiratory failure among COVID-19 occurs in 42% of patients with COVID-19 pneumonia, and 61-81% of patients requiring intensive care . Among the suggested treatments for the management of ARDS patients, prone position (PP) can be used as an adjuvant therapy for improving ventilation in these patients, as recommended in the Surviving Sepsis Campaign COVID-19 guidelines. Nevertheless, no data is currently available on application and feasibility of PP in invasively ventilated patients with COVID-19 on their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed COVID-19 infection
* Prone positioning in patients admitted to ICU undergoing invasive Mechanical Ventilation

Exclusion Criteria:

* Bedsides contraindications to the Prone Positioning and patients in PP but undergoing Non- invasive ventilation should be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All critically ill patients undergoing PP in the enrolling centers will be retrospectively and prospectively observed.
  It should be underlined that the lack of consensus concerning the timing and duration of PP leads to variability in clinical practice and treatments are initiated in accordance with the judgement of the responsible physician. Under these circumstances, it is preferable to keep web-based, multicenter, observational registry" inclusion criteria as wide as possible so as to obtain a real picture of the clinical practice worldwide.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the subpopulation of critically ill patients that most benefits from prone positioning their intermediate surrogate endpoints. Identification of the subpopulation of critically ill patients with COVID-19 that most benefits from | through study completion, an average of 1 year
  This subpopulation will be described using the baseline variables associated with a positive long-term patient's outcome. In particular baseline variables statistically associated through multivariable regression analyses with the patient's survival at hospital discharge will be identified and expressed with their Odds ratios, 95%CI and p-value

SECONDARY OUTCOMES:
Description of the over-time variation of clinical variables during prone positioning | through study completion, an average of 1 year
  this over-time variation will be expressed, for each variable, as a percentage variation compared with the baseline value (at the prone position initiation).static compliance of the respiratoty system will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Silvia De Rosa, Principal Investigator — Ospedale San Bortolo di Vicenza
Locations (1):
- Silvia De Rosa, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lucchini A, Bambi S, Mattiussi E, Elli S, Villa L, Bondi H, Rona R, Fumagalli R, Foti G. Prone Position in Acute Respiratory Distress Syndrome Patients: A Retrospective Analysis of Complications. Dimens Crit Care Nurs. 2020 Jan/Feb;39(1):39-46. doi: 10.1097/DCC.0000000000000393. PMID 31789984
- [Result] Carsetti A, Damia Paciarini A, Marini B, Pantanetti S, Adrario E, Donati A. Prolonged prone position ventilation for SARS-CoV-2 patients is feasible and effective. Crit Care. 2020 May 15;24(1):225. doi: 10.1186/s13054-020-02956-w. No abstract available. PMID 32414420
- [Result] Coppo A, Bellani G, Winterton D, Di Pierro M, Soria A, Faverio P, Cairo M, Mori S, Messinesi G, Contro E, Bonfanti P, Benini A, Valsecchi MG, Antolini L, Foti G. Feasibility and physiological effects of prone positioning in non-intubated patients with acute respiratory failure due to COVID-19 (PRON-COVID): a prospective cohort study. Lancet Respir Med. 2020 Aug;8(8):765-774. doi: 10.1016/S2213-2600(20)30268-X. Epub 2020 Jun 19. PMID 32569585
- [Derived] De Rosa S, Sella N, Rezoagli E, Lorenzoni G, Gregori D, Bellani G, Foti G, Pettenuzzo T, Baratto F, Fullin G, Papaccio F, Peta M, Poole D, Toffoletto F, Maggiore SM, Navalesi P; SIAARTI Study Group. The PROVENT-C19 registry: A study protocol for international multicenter SIAARTI registry on the use of prone positioning in mechanically ventilated patients with COVID-19 ARDS. PLoS One. 2022 Dec 30;17(12):e0276261. doi: 10.1371/journal.pone.0276261. eCollection 2022. PMID 36584022
- See also: Related Info — https://www.siaarti.it/news/418384